CLINICAL TRIAL: NCT02209285
Title: Self-Management Program for Older Adults With Multimorbidity: A Pragmatic Randomized Controlled Trial
Brief Title: Self-Management Program for Older Adults With Multimorbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Maureen Markle-Reid, Professor and Canada Research Chair, Co-Scientific Director of Aging, Community and Health Research Unit (ACHRU), McMaster University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: STRCT- 06669
Record Dates: First submitted 2014-07-07; First posted 2014-08-05 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Multimorbidity
Keywords: Older adults; Home and community care; Effectiveness; Cost analysis; Pragmatic trial; Self-management
MeSH Terms: interventions — Self-Management; Aging; Multimorbidity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): The control group will receive usual care, which is provided by the community care access centre (CCAC). Usual care may include in-home visits by regulated health care providers, personal support workers, and care coordination through the community care access centre. Case conferences may occur on an as-needed basis.
- Self-Management Program for Older Adults with Multimorbidity (Active Comparator): Individuals in the intervention group will receive a six-month self-management intervention consisting of three components: (1) intensive case management and community navigation; (2) a maximum of two in-home visits by the care coordinator, two in-home visits by a Registered Nurse, and three in-home visits by the Occupational therapist or Physiotherapist, and six visits by a Personal Support Worker over 6 months in addition to usual home care services; and (3) monthly interprofessional team case conferences to develop an evidence-based, patient-centred community reintegration plan.
  Interventions: Behavioral: Self-Management Program for Older Adults with Multimorbidity

INTERVENTIONS:
Behavioral: Self-Management Program for Older Adults with Multimorbidity — Individuals in the intervention group will receive a six-month community intervention consisting of three components: (1) intensive case management and community navigation; (2) a maximum of two in-home visits by the care coordinator, two in-home visits by a Registered Nurse, and three in-home visits by the Occupational therapist or Physiotherapist, and six visits by a Personal Support Worker over 6 months in addition to usual home care services; and (3) monthly interprofessional team case conferences to develop an evidence-based, patient-centred community reintegration plan.
  Arms: Self-Management Program for Older Adults with Multimorbidity

SUMMARY:
Patients with multimorbidity move between multiple care settings, and so they are at high risk of receiving fragmented care leading to increased risk for avoidable illness, death, and health care costs. Recent Canadian studies and reports identify significant gaps in the delivery of effective care to patients with multiple chronic conditions in community-based settings.

The overall goal of the intervention is to promote successful management of chronic conditions, enhance quality of life, reduce the on-demand use of expensive health services and support primary caregivers (i.e. family or friends) who provide physical, emotional or financial care to an older adult with multimorbidity. This research program will leverage the tremendous potential to reduce the burden of multimorbidity by enhancing community-based prevention and chronic disease management.

This pragmatic mixed-methods randomized controlled trial will evaluate the effectiveness of an interprofessional team-based self-management intervention on health-related quality of life (HRQOL), depression, anxiety, self-efficacy, and the costs of use of health services for older adults with multimorbidity receiving home care and their family caregivers. The results will inform: (1) the development of national standards for community-based care for patients with multimorbidity and (2) the development of a new and innovative community-based model for the management of multimorbidity that can be scaled up and spread across Canada.

DETAILED DESCRIPTION:
Research Question:

What is the acceptability and effects of a six-month self-management program compared to usual home care services for older adults with multimorbidity and their family and friend caregivers?

Methods:

The design is a pragmatic, mixed-methods; randomized controlled trial with individuals newly referred to and using home care services. The intervention is a 6-month self-management program for older adults with multimorbidity. It will be provided by an interprofessional team of home care providers and will consist of three components: (1) intensive case management to facilitate access to services across the care continuum, provide psychosocial support and advocacy, and coordinate home care; (2) a minimum of two in-home visits by the Community Care Access Centre (CCAC) Case Manager, two visits by the Registered Nurse (RN), three visits by the Physiotherapist (PT) or Occupational Therapist (OT), and six visits by a Personal Support Worker (PSW) over 6 months in addition to usual home care services. The in-home visit schedule and team composition will be tailored to client needs and will be determined in collaboration with the home care providers. The interprofessional (IP) team will conduct comprehensive screening and assessments for chronic conditions, utilize strengths-based practice to encourage self-management and foster behavioural change, provide education for multimorbidity, medication review and management, in-home exercise, and caregiver support; and (3) monthly interprofessional team case conferences to develop an IP evidence-based, patient-centred care plan.

Outcomes will be assessed at baseline and 6 months. Summary descriptive measures will be reported for all variables. Analysis of covariance will be used to compare study groups, while adjusting for baseline measurements and potential confounding variables. Subgroup analyses will be conducted based on sex/gender and region.

Expected Outcomes:

It is expected that older adults receiving the intervention will show greater improvements in health-related quality of life compared to usual home care services. These improvements will be achieved at no additional cost, from a societal perspective.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age and older;
* Three or more chronic conditions
* Newly referred (following initiation of the study) for home care services and living in the community, including supportive housing, retirement homes, and lodging homes and excluding long-term care;
* Able to speak English or have access to a translator;
* Not planning to move away from the CCAC catchment area in the next 6 months;
* Be mentally competent to provide informed consent, either independently or by a substitute decision maker.

Exclusion Criteria:

* Participants will be excluded if they are unable to read and understand English and do not have access to their own translator

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Physical Component Summary Score of the Short-Form 12 Health Survey, Version 2 (SF-12v2) | Baseline and end of study (6 months from baseline)
  The Short-Form 12 Health Survey will be administered to older adult participants to measure health-related quality of life.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder Screener (GAD-7) Scale | Baseline and end of study (6 months from baseline)
  The GAD-7 will be administered to older adult participants at baseline and 6 months to assess anxiety.
Health and Social Services Utilization Inventory (HSSUI) | Baseline and end of study (6 months from baseline)
  The HSSUI will be administered to older adult participants at baseline and 6 months to assess healthcare utilization costs.
Centre for Epidemiological Studies in Depression - Shortened version (CES-D-10) | Baseline and end of study (6 months from baseline)
  The CES-D-10 will be administered to older adult participants at baseline and 6 months to assess depressive symptoms
  It is estimated that approximately 70% of the study participants will have a family caregiver.
Collaborative Practice Assessment Tool (CPAT) | At 3 months and at 9 months after the start of the study
  The CPAT will be administered to participating home care providers at 3 months and 9 months after initiation of the intervention to assess changes in collaborative practice.
Mental Component Summary Score of the Short-Form 12 Health Survey, Version 2 (SF-12v2) | Baseline and end of study (6 months from baseline)
  The Short-Form 12 Health Survey will be administered to older adult participants to measure health-related quality of life.
Self-efficacy for managing chronic disease scale | Baseline and end of study (6 months from baseline)
  The self-efficacy for managing chronic disease scale will be administered to older adult participants to assess their level of self-efficacy
Team Climate Inventory-19 (TCI-19) | At 3 months and at 9 months after the start of the study
  The TCI-19 will be administered to participating home care providers at 3 months and 9 months after initiation of the intervention to assess the level of team functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Markle-Reid, RN, PhD, Principal Investigator — McMaster University, School of Nursing; Jenny Ploeg, RN, PhD, Principal Investigator — McMaster University, School of Nursing
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Markle-Reid M, Ploeg J, Valaitis R, Duggleby W, Fisher K, Fraser K, Ganann R, Griffith LE, Gruneir A, McAiney C, Williams A. Protocol for a program of research from the Aging, Community and Health Research Unit: Promoting optimal aging at home for older adults with multimorbidity. J Comorb. 2018 Jul 31;8(1):2235042X18789508. doi: 10.1177/2235042X18789508. eCollection 2018. PMID 30191144